CLINICAL TRIAL: NCT02669316
Title: Adherence to Mediterranean Diet and Physical Exercise Profile in NAFLD: Relationship With Echocardiography Measures in Non-diabetic Subjects.
Brief Title: Echocardiography, Adherence to Mediterranean Diet (AMDS) and Physical Exercise in Fatty Liver
Acronym: CARDIONAFLD
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera, Universitaria Policlinico Vittorio Emanuele (Other)
Responsible Party: Principal Investigator, Guglielmo Trovato, MD, PhD, Dirigente Medico, Azienda Ospedaliera, Universitaria Policlinico Vittorio Emanuele
Other Study IDs: CARDIONAFLD
Record Dates: First submitted 2016-01-18; First posted 2016-02-01 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Fatty Liver
Keywords: diet
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
NAFLD is associated with unhealthy lifestyle and obesity, without alcohol habits. An association of NAFLD with coronary artery disease and with impaired heart function was reported, but without considering severity of NAFLD and with the bias of including diabetes. Aim: to challenge if severity of liver steatosis assessed by UltraSound Bright Liver Score (BLS) can predict the impairment of systolic heart function, assessed by echocardiography (Ejection Fraction, EF), diastolic function (assessed by E/A ratio), Left Ventricular Mass, Left atrial diameter.

DETAILED DESCRIPTION:
METHOD and measures: Age, obesity (BMI) , dietary profile (assessed as Adherence to Mediterranean Diet Score, AMDS), physical activity profile, assessed by the Baecke's physical exercise questionnaire, Insulin resistance (assessed by HOMA) were all taken into account for their confounding and synergic effect. Multiple regression analysis and Odds ratio will be the statistical tools that will be used.Receiver operator curve (ROC) analysis will be applied in order to find the cut-off, if any, of the considered measures vs. NAFLD and significant abnormalities of echocardiography measures.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis on fatty liver

Exclusion Criteria:

* Diabetes
* Cancer
* virus hepatitis
* alcohol habits above 20 g/day (140 g/week) and any binge drinking
* myocardial infarction,
* valvular or congenital heart disease
* heart failure
* respiratory or renal insufficiency
* rheumatic or autoimmune disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects withour acute or chronic disease checked by US imaging of the liver during routine work-up for dietary and physical exercise counseling
Sampling Method: Non-Probability Sample
Enrollment: 660 (Actual)
Dates: Start 2008-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Left Ventricular Myocardial mass: the measurement described below is echo-cardiographic, taken according to the joint guidelines of the American and European Societies of Echocardiography with appropriate equipments. | through study completion, an average of 4 years
  left ventricular mass indexed by body surface area g/m2.

SECONDARY OUTCOMES:
assessment of diastolic function: the measurement described below is echo-cardiographic, taken according to the joint guidelines of the American and European Societies of Echocardiography with appropriate equipments. | through study completion, an average of 4 years
  Doppler transmitral E/A ratio
assessment of systolic function: the measurement described below is echo-cardiographic, taken according to the joint guidelines of the American and European Societies of Echocardiography with appropriate equipments. | through study completion, an average of 4 years
  ejection fraction (%)

CONTACTS AND LOCATIONS:
Overall Officials: GUGLIELMO TROVATO, MD, Principal Investigator — University of Catania - Policlinico
Locations (1):
- Guglielmo Trovato, Catania, CT, Italy

IPD SHARING:
Plan to Share IPD: No